CLINICAL TRIAL: NCT05099354
Title: The Effect of Endovascular Thrombectomy on Autonomic Nervous System in Patients With Large-vessel Ischemic Stroke - a Prospective Descriptive Pilot Study (AFFRICATE)
Brief Title: The Effect of Endovascular Thrombectomy on Autonomic Nervous System in Patients With Large-vessel Ischemic Stroke
Acronym: AFFRICATE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Karl Landsteiner University of Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: AFFRICATEThrombectomy
Record Dates: First submitted 2021-09-08; First posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Autonomic Nervous System
Keywords: stroke; thrombectomy; autonomic nervous system
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: autonomic nervous system testing — * Autonomic tests, including heart rate variability (HRV) and baroreceptor sensitivity (BRS), are performed with a 10min ECG with non-invasive or invasive blood pressor measuring during rest. During the time at the stroke unit, this data will be calculated using the existing continuous monitoring.
  * Valsalva maneuver during continuous ECG and blood pressure monitoring. The patient will be instructed to exhale against a mouthpiece with a defined resistance for 15 seconds.
  * Assessment of the cerebrovascular reserve capacity will be done with continuous transcranial duplex sonography (TCD) and "breath holding index" (BHI). The patient will be instructed to hold his breath for 30 seconds, 4 times in a row with intervals of 4 minutes. This test will be performed only in responsive and compliant patients.

SUMMARY:
The autonomic nervous system (ANS), regulating involuntary physiologic processes including heart rate and blood pressure, is affected by changes in the cerebral vessels like carotid artery stenosis, occlusion, carotid artery stent and endarterectomy.

Until now, no data concerning autonomic nervous system in patients with acute intracranial large artery occlusion and thrombectomy is available. Due to the known effect on ANS in case of pathologies of extracranial brain supplying arteries it is highly suspected that intracranial large artery occlusion and thrombectomy can affect the ANS as well.

The aim of this project is to determine autonomic parameters during and after thrombectomy in patients with large cerebral artery occlusion. The project is a prospective descriptive pilot study at the University Hospital Tulln. 20 patients will be assessed during and after thrombectomy up to three months post intervention. A combination of autonomic parameters, hemodynamic parameters and clinical outcome will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age: > 18 years of age
* Acute ischemic stroke with large extra- and intracranial artery occlusion and intraarterial mechanical thrombectomy treatment.
* Successful recanalization after thrombectomy with TICI 2b or 3.
* Informed consent by the patient

Exclusion Criteria:

* Informed consent not possible within 7 days after thrombectomy due to impaired awareness or speech disturbances.
* Permanent stent during thrombectomy.
* Severe complications, such as severe intracranial hemorrhage, during or after thrombectomy including prolonged ICU stay.
* Modified rankin scale (mRS) over 3 before admission.
* Diagnosis of dementia with mini mental state examination (MMSE) < 26 points in the medical history
* Intracranial hypertension in the medical history or brain imaging.
* Patent foramen ovale in the medical history.
* Glaucoma in medical history.
* Inability to complete study visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 patients treated with thrombectomy at the University Hospital Tulln during a period of 12 months, meeting inclusion and exclusion criteria will be included in the study.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
heart rate variability | change in baseline after 3 months
  heart rate variability measured by 30 minute continuous ecg
baro receptor sensitivity | change in baseline after 3 months
  calculated from continuous ecg and continuous non-invasive blood pressure over 30 minutes

IPD SHARING:
Plan to Share IPD: No